CLINICAL TRIAL: NCT03738124
Title: Evaluation of the Valiant Mona LSA Thoracic Stent Graft System in Thoracic Aortic Aneurysms and Chronic Dissections
Acronym: MONA-LSA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Production of the medical device was stopped
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: RC31/18/0234
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Aortic Aneurysm, Thoracic
Keywords: stent graft; branch stent graft; thoracic aneurysm; endovascular aortic repair; aortic dissection; Valiant Mona LSA Thoracic Stent Graft System
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Valiant Mona LSA Thoracic Stent Graft System (Experimental): The Valiant Mona LSA Thoracic Stent Graft System is administered.
  Interventions: Device: Valiant Mona LSA Thoracic Stent Graft System

INTERVENTIONS:
Device: Valiant Mona LSA Thoracic Stent Graft System — The Valiant Mona LSA device is a modular two-component system consisting of a main stent graft (MSG) and a branch stent graft (BSG), delivered separately, designed to maintain LSA perfusion. Briefly, under general anesthesia and after heparin injection, a MSG access is achieved via a femoral artery. A Through-and-through wire access for delivery of the BSG is achieved via a brachial artery. After the placement of the main aortic stent graft in the arch with the cuff at the level of the ostium of the LSA, the BSG is placed through a femoral access.

SUMMARY:
To ensure adequate seal of currently available stent grafts, a proximal 20 mm of healthy aorta is recommended. Extending the proximal landing zone into the arch by intentional covering of the left subclavian artery (LSA) without revascularization expose to serious neurologic complications. Serious risks are also known to accompany subclavian revascularization. The Valiant Mona LSA Thoracic Stent Graft System (Medtronic,Santa Rosa, Calif) consists of a main stent graft and a branch stent graft designed to maintain LSA patency. The purpose of this study is to characterize the safety and effectiveness of this device for the treatment of Aneurysms and chronic Type B dissections of the arch.

DETAILED DESCRIPTION:
Stent graft coverage of the left subclavian artery (LSA) may be required to achieve an adequate landing zone in up to 40% of descending thoracic aneurysms (DTAs). To ensure adequate seal of currently available off-the-shelf stent grafts, 20 mm of healthy aorta is recommended between the proximal neck of the aneurysm and the leading edge of the stent graft. Stent graft placement can be facilitated by extending the proximal landing zone into the arch and covering the LSA; however, there may be a higher risk of serious neurologic outcomes (cerebral and paraplegia), although this is still a matter of debate. Serious risks are also known to accompany subclavian revascularization, which may involve bypass or transposition. The Valiant Mona LSA Thoracic Stent Graft System (Medtronic,Santa Rosa, Calif) consists of a main stent graft and a branch stent graft designed to maintain LSA patency while diverting circulation through the encroaching aneurysm.

The purpose of the feasibility study is to characterize the safety of the Valiant Mona LSA Thoracic Stent Graft System, including an assessment of the safety and effectiveness of the device acutely and at the 1-month visit in the identified subject population (Aneurysms and chronic, Type B dissections). A follow up of this population will be annually during 5 years.

This pilot, non-randomized, single-arm prospective study will concern 20 patients. Inclusion criteria required patients with a thoracic aortic aneurysm (TAA) or dissection with an indication of a stent-Graft insertion. Primary end points will be aneurysm-related mortality, stroke, paraplegia, left arm/hand ischemia, and treatment success. Technical success will be assessed by imaging at 1 month, 6 months then annually during 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age.
* Subject understands and has signed an Informed Consent
* Subject must be considered a candidate for revascularization of the LSA.
* Subject must be able to tolerate a surgical revascularization of the LSA.
* Subject has a descending thoracic aneurysm (DTA) which will require coverage of the LSA
* Subject has a healthy, non-diseased aortic proximal seal zone of at least 10 mm from the left carotid to the LSA and at least 5 mm landing zone distal to the LSA and proximal to the start of the aneurysm/ulcer/or the proximal entry tear for dissection.
* Subject has a non-diseased aortic diameter between 25 mm and 42 mm (fusiform/saccular aneurysms or penetrating ulcers) or 28 mm to 44 mm (chronic type B dissections),
* Subject has a LSA with a diameter between 8 mm and 13 mm.
* Subject has sufficient landing zone within the LSA to accommodate the BSG without occlusion of any significant vessels
* Subject has patent brachial arteries, iliac or femoral arteries (without circumferential calcifications and a diameter of ≥ 10mm), or can tolerate a conduit that will allow endovascular access to the aneurysmal site with the delivery system of the appropriate sized device chosen for treatment.
* Subject has a condition requiring prospective revascularization of the LSA

Exclusion Criteria:

* Subject has an aneurysmal, tortuous, or atherosclerotic LSA, conflicting the branch graft insertion.
* Subject has an aortic atheroma classified as grade IV or grade V.
* Subject has prohibitive calcification, occlusive disease, or tortuosity of intended fixation sites.
* Treatment with the Valiant Mona LSA Thoracic Stent Graft system would require intentional coverage of the left common carotid artery with the stent graft fabric.
* Subject has significant and/or circumferential aortic mural thrombus at either the proximal or distal attachment sites that would compromise fixation and seal of the device.
* Subject is a pregnant or breastfeeding female.
* Subject has a known allergy or intolerance to the device components.
* Subject is in acute renal failure or has renal insufficiency with a serum creatinine ≥ 2.0 mg/dL or is on dialysis.
* Subject has coronary artery disease with unstable angina and has not received treatment.
* Subject has a connective tissue disease (e.g. Marfan's syndrome, medial degeneration).
* Subject has active systemic infection and/or a mycotic aneurysm.
* Subject is currently participating in an investigational drug or device clinical trial that would interfere with the observations of this study.
* Subject has other medical, social, or psychological problems that, in the opinion of the investigator, will interfere with treatment and follow-up procedures.
* Subject has a life expectancy of less than 1 year.
* Subject has a history of bleeding diathesis, coagulopathy, or refuses blood transfusion.
* Subject has a known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Safety events (aorta related mortality, stroke, paraplegia, left arm/hand ischemia) | 1 month
  Composite endpoint defined as the occurrence of one of the following events: aorta related mortality, stroke, paraplegia, left arm/hand ischemia
Effectiveness | 1 month
  Effectiveness defined as technical success and successful exclusion of the aneurysm or false lumen while maintaining patency of the main stent graft (MSG) and branch stent graft (BSG)

SECONDARY OUTCOMES:
Aorta related mortality | 6 months, 12 months, 24 months, 36 months, 48 months and 60 months
  Occurrence of aorta related mortality
Stroke | 6 months, 12 months, 24 months, 36 months, 48 months and 60 months
  Occurrence of stroke
Paraplegia | 6 months, 12 months, 24 months, 36 months, 48 months and 60 months
  Occurrence of paraplegia
Left arm/hand ischemia | 6 months, 12 months, 24 months, 36 months, 48 months and 60 months
  Occurrence of left arm/hand ischemia
Effectiveness (Successful exclusion of the aneurysm) | 6 months, 12 months, 24 months, 36 months, 48 months and 60 months
  Successful exclusion of the aneurysm
Effectiveness (patency) | 6 months, 12 months, 24 months, 36 months, 48 months and 60 months
  False lumen while maintaining patency of the main stent graft (MSG) and branch stent graft (BSG)
Duration of the intervention | Day 0
  Duration of the intervention
Necessary time for the branch placement | Day 0
  Necessary time for the branch placement
Characteristics of the intervention (general anaesthesia) | Day 0
  General anaesthesia performing
Characteristics of the intervention (blood loss) | Day 0
  Blood loss volume
Characteristics of the intervention (transfusion) | Day 0
  Transfusion performing
Duration of the stay in intensive care | Day 0
  Duration of the stay in intensive care
Duration of the hospitalization | Day 0
  Duration of the hospitalization
Characteristics of the hospitalization (intraoperative complications) | Day 0
  Occurrence of intraoperative complications
Quality of life with EuroQol-5D | Baseline, 6 months, 12 months, 24 months, 36 months, 48 months and 60 months
  The quality of life will be measured with the EuroQol-5D (5 levels) questionnaire
Minor adverse events | 1 month, 6 months, 12 months, 24 months, 36 months, 48 months and 60 months
  Occurrence of minor adverse events
Serious adverse events | 1 month, 6 months, 12 months, 24 months, 36 months, 48 months and 60 months
  Occurrence of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hervé ROUSSEAU, MD, Principal Investigator — University Hospital of Toulouse
Locations (2):
- France (2):
  - Hôpital Timone Adultes, Marseille
  - CHU Toulouse, Hôpital Rangueil, Toulouse

IPD SHARING:
Plan to Share IPD: No